CLINICAL TRIAL: NCT03547830
Title: A Clinical Trial of Plerixafor With G-CSF as Additional Agents in Conditioning Regimen for Prevention of Graft Failure in Patients With Chronic Granulomatous Disease
Brief Title: Plerixafor/G-CSF as Additional Agents for Conditioning Before HSCT in CGD Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2018-02
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Granulomatous Disease
Keywords: chronic granulomatous disease; graft failure; stem cell transplantation; plerixafor; conditioning regimen
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plerixafor/G-CSF (Experimental): Plerixafor/G-CSF for HSCT conditioning Myeloablative conditioning regimen with Plerixafor as addition agent before stem cell transplantation in CGD patients
  Interventions: Drug: Plerixafor; Drug: Gcsf

INTERVENTIONS:
Drug: Plerixafor — Plerixafor for Conditioning before HSCT.
Drug: Gcsf — GCSF for Conditioning before HSCT.

SUMMARY:
Treatment Study to assess of safety and efficiency of conditioning with Plerixafor and G-CSF as additional agents for prevention of graft failure after transplantation in patients with chronic granulomatous disease

DETAILED DESCRIPTION:
Severe primary or secondary graft dysfunction is one of major problem in patients with Chronic granulomatous disease (CGD). In this study the hypothesis is that the use of plerixafor and G-CSF as additional agents in conditioning regimen would offers advantages. The effect is based on mobilizing bone marrow stem cells into the peripheral blood and blocking CXCR4 chemokine receptors to prevent stem cell homing. Thus, some have hypothesized that plerixafor and G-CSF make free stromal space of the bone marrow available for donor stem cell engraftment. Moreover, stem cell release probably leads to liberation of host stem cells from the anti-apoptotic effects of the BM stroma for the more powerful effect of chemotherapy. Thus, the purpose of this study is to evaluate the safety and efficiency of myeloablative conditioning with Plerixafor and G-CSF as additional agents for prevention of graft failure after stem cell transplantation in patients with chronic granulomatous disease.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 1 months and < 25 years Patients diagnosed with CGD eligible for an allogeneic transplantation Signed written informed consent

Exclusion Criteria:

Lack of informed consent.

Ages: 1 Month to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Estimated)
Dates: Start 2019-04-13 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 1 year
  The EFS probability compared with historical control. We mean event as primary (non-engraftment) and secondary (rejection) graft dysfunction.

SECONDARY OUTCOMES:
1. Overall survival | 1 year
  The OS probability compared with historical control
Proportion of patients with full/mixed donor chimerism | 30 days
  Evaluation of the percentage of patients with the full/mixed donor chimerism (whole blood and CD3+ lineage). In addition, patients will be divided in accordance with % of donors cells: >95%; 50%-95%; 10%-49%; <10%. All data will be compared with historical control
3. Transplant related mortality | 1 year
  The TRM probability compared with historical control.
4. Acute Graft Versus Host Diseases | 100 days
  Cumulative Incidence of aGVHD
5. Incidence of Plerixafor related toxicity | 100 days
  severity, features, incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Background] Balashov D, Laberko A, Shcherbina A, Trakhtman P, Abramov D, Gutovskaya E, Kozlovskaya S, Shelikhova L, Novichkova G, Maschan M, Rumiantsev A, Maschan A. A Conditioning Regimen with Plerixafor Is Safe and Improves the Outcome of TCRalphabeta+ and CD19+ Cell-Depleted Stem Cell Transplantation in Patients with Wiskott-Aldrich Syndrome. Biol Blood Marrow Transplant. 2018 Jul;24(7):1432-1440. doi: 10.1016/j.bbmt.2018.03.006. Epub 2018 Mar 14. PMID 29550630